CLINICAL TRIAL: NCT03601221
Title: Observational Study on Seroprevalence of Hepatitis E Infection in Healthy Blood Donors in the Canton Ticino
Brief Title: Seroprevalence Hepatitis E Infection in Healthy Blood Donors
Status: Completed | Type: Observational
Sponsor: Ente Ospedaliero Cantonale, Bellinzona (Other)
Collaborators: Swiss Transfusion SRC (Other); Clinical Trial Unit Ente Ospedaliero Cantonale (Other)
Responsible Party: Sponsor
Other Study IDs: HEV-TI-2018
Record Dates: First submitted 2018-07-05; First posted 2018-07-26 (Actual); Last update posted 2020-03-31 (Actual); Status verified 2020-03

CONDITIONS: Hepatitis E
MeSH Terms: conditions — Hepatitis E | interventions — Specimen Handling

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Sample collection — Collection of one sampling pouch from each blood donor

SUMMARY:
This is a HEV seroprevalence in the health donors in the Canton Ticino study. The pre-donation sampling pouch of each blood donor coming form the Cantone Ticino region will be collected and tested for HEV serology (IgM and IgG).

DETAILED DESCRIPTION:
Pre-donation sampling pouch of fresh and stored frozen plasma collected within the last 5 years will be tested for HEV IgG serology at the National Reference Laboratory of the Blood Transfusion Services SRC in Berne Collected data will be used to determine HEV seroprevalence, actual and in the last 5 years, in the Canton Ticino and to investigate trend and pattern of the HEV infection (seroprevalence by different regional areas, comparison with national HEV data, and correlation with age, sex and place of residence).

ELIGIBILITY:
Inclusion Criteria:

* Healthy and voluntary blood donors
* Subjects living in the Canton Ticino
* Inclusion criteria for blood donation
* Signed informed consent of the STCRS SI for blood donation

Exclusion Criteria:

* Exclusion criteria for blood donation

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Healthy and voluntary blood donors
Sampling Method: Non-Probability Sample
Enrollment: 1447 (Actual)
Dates: Start 2018-05-29 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
HEV blood incidence | One year
  HEV incidence assessed through a single periferal blood sample from each donor

SECONDARY OUTCOMES:
change in the blood incidence of HEV | Five years
  Determine the change in the incidence of HEV in the Canton Ticino region in the last 5 years analysing the blood sample of the donors.
Geogarphical distribution of the HEV measured in the blood sample | Five years
  Determination of the distribution of the HEV infection in different geographical areas of the Canton Ticino analysing donor blood samples
Trend of the HEV infection measured in the blood sample | One year
  Evaluation of the trend of the HEV infection in the CantoneTicino compared to other Swiss cantons

CONTACTS AND LOCATIONS:
Overall Officials: Florian Bihl, MD, Study Director — Ente Ospedaliero Cantonale, Bellinzona
Locations (1):
- Swiss Transfusion SRC Canton Ticino, Lugano, Switzerland

IPD SHARING:
Plan to Share IPD: No